CLINICAL TRIAL: NCT01679665
Title: Systems Biology of Vaccination for EV71 Vaccine in Chinese Healthy Children Aged From 2 to 5 Years Old
Brief Title: Systems Biology of Vaccination for EV71 Vaccine in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Bejing Vigoo Biological Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT012
Record Dates: First submitted 2012-09-01; First posted 2012-09-06 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Systems Biology; Early Gene; EV71 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 320U /0.5ml in children (from 2 to 5 years old) (Experimental): inactivated vaccine(vero cell) against EV71 of 320U /0.5ml in 48 children aged 2-5 years old on day 0,28
  Interventions: Biological: 320U /0.5ml
- 0/0.5ml placebo in children (from 2 to 5 years old) (Placebo Comparator): 0/0.5ml placebo in 24 children aged 2-5 years old on day 0, 28
  Interventions: Biological: 0/0.5ml placebo

INTERVENTIONS:
Biological: 320U /0.5ml — inactivated vaccine(vero cell) against EV71 of 320U /0.5ml, two doses, 4 weeks interval
  Arms: 320U /0.5ml in children (from 2 to 5 years old)
Biological: 0/0.5ml placebo — 0/0.5ml placebo, two doses, 4 weeks interval
  Arms: 0/0.5ml placebo in children (from 2 to 5 years old)

SUMMARY:
Recently, an inactivated vaccine (vero cell) against EV71 has been investigated in Phase 1 and Phase 2 clinical trials. Data from these trials showed that the EV71 vaccine has good safety profile and was immunogenic. 320 U alum-adjuvant vaccine has been chosen as the candidate vaccine for the phase 3 clinical trial.

This clinical trial is a supplementary phase 2 trial, which is designed to study the gene expression patterns induced by EV71 vaccine in Chinese healthy children aged from 2 to 5 years old use a systems biology approach combined with microarray analysis，RT-PCR and neutralizing antibody testing for PBMC and serum collected form the studied children population, to predict immunogenicity, and explore mechanistic insights about the EV71 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged from 2 to 5 years old as established by medical history and clinical examination
* The pre-vaccination neutralizing antibody against EV71 <1:8 which is determined by ELISA
* The subjects' guardians are able to understand and sign the informed consent
* Had never received the vaccine against EV71
* Subjects who can and will comply with the requirements of the protocol
* Subjects with temperature <37.1°C on axillary setting

Exclusion Criteria:

* Subject who has a medical history of HFMD
* <= 37 weeks gestation
* Subjects with a birth weight <2.5 kg
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine
* Family history of seizures or progressive neurological disease
* Family history of congenital or hereditary immunodeficiency
* Severe malnutrition or dysgenopathy
* Major congenital defects or serious chronic illness, including perinatal brain damage
* Autoimmune disease
* Bleeding disorder diagnosed by a doctor or significant bruising or bleeding difficulties with IM injections or blood draws
* Any acute infections in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6month
* Any prior administration of blood products in last 3 month
* Any prior administration of other research medicines in last 1month
* Any prior administration of attenuated live vaccine in last 28 days
* Any prior administration of inactivated vaccines in last 14 days, such as pneumococcal vaccine
* Under the anti - TB prevention or therapy
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Genomic signatures that predicted immune responses in infants vaccinated with EV71 vaccine | Frame: 3 days after first dose
  Identifying genomic signatures that predicted immune responses in infants vaccinated with EV71 vaccine at day 3 in children aged 2-5 years
Genomic signatures that predicted immune responses in infants vaccinated with EV71 vaccine | 7 days after first dose
  Identifying genomic signatures that predicted immune responses in infants vaccinated with EV71 vaccine at day 7 in children aged 2-5 years
Genomic signatures that predicted immune responses in infants vaccinated with EV71 vaccine | 28 days after first dose
  Identifying genomic signatures that predicted immune responses in infants vaccinated with EV71 vaccine at day 28 in children aged 2-5 years
Genomic signatures that predicted immune responses in infants vaccinated with EV71 vaccine | 28 days after second dose
  Identifying genomic signatures that predicted immune responses in infants vaccinated with EV71 vaccine at day 56 in children aged 2-5 years
Genomic signatures that predicted immune responses in infants vaccinated with EV71 vaccine | 6 months after first dose
  Identifying genomic signatures that predicted immune responses in infants vaccinated with EV71 vaccine at month 6 in children aged 2-5 years

SECONDARY OUTCOMES:
GMT, seroconversion rate of anti-EV71 antibodies in serum after first vaccination | 28 days after the first vaccination
  GMT, seroconversion rate of anti-EV71 antibodies in serum 28 days after first vaccination
GMT, seroconversion rate of anti-EV71 antibodies in serum after second vaccination | 28 days after second vaccination
  GMT, seroconversion rate of anti-EV71 antibodies in serum 28 days after second vaccination
the safety of EV71 vaccine in healthy children aged 2-5 years | 28 days after the first dose
  Frequency of systemic and local adverse reactions within 28 days after the first dose of EV71 vaccine in healthy children aged 2-5 years
the safety of EV71 vaccine in healthy children aged 2-5 years | 28 days after the second dose
  Frequency of systemic and local adverse reactions within 28 days after the second dose of EV71 vaccine in healthy children aged 2-5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China